CLINICAL TRIAL: NCT06314451
Title: Cross-condition Validation of the Patient Reported Outcome Measure for Patients Receiving Glucocorticoids (the Steroid PRO)
Brief Title: Cross-condition Validation of the Steroid PRO
Status: Recruiting | Type: Observational
Sponsor: University of the West of England (Other)
Collaborators: Johns Hopkins University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: HAS.22.11.035
Record Dates: First submitted 2023-03-16; First posted 2024-03-18 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Disease; Immune System Disorder; Gastrointestinal Diseases; Dermatologic Disease; Respiratory Disease
Keywords: Glucocorticoids; Steroids; Health-related quality of life; Rheumatology; Respiratory; Gastroenterology; Dermatology; Pulmonology; Patient; Patient reported outcomes
MeSH Terms: conditions — Immune System Diseases; Gastrointestinal Diseases; Skin Diseases; Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with respiratory, gastroenterology and dermatology inflammatory conditions: Patients will be purposively sampled to include a spectrum of participants with a range of different diseases and demographics (age, gender, country) for each indication. Sample size will also be led by the point at which no further issues are emerging during the cognitive interview process.
  Interventions: Other: Cognitive Interview
- Clinicians and researchers skilled in inflammatory diseases: Clinician researchers from each country (UK, USA) will be purposively sampled to include a spectrum of participants with a range of clinical experience and demographics (age, gender, country). Sample size will also be led by the point at which no further issues are emerging during the cognitive interview process.
  Interventions: Other: Cognitive Interview

INTERVENTIONS:
Other: Cognitive Interview — The study involves a single cognitive interview with a researcher, either online, by telephone, or face-to-face. People who want to take part will be given information about the study and asked to give written consent. Then they will be asked to talk about the wording of the questionnaire and how relevant it is to them.
  Cognitive interviewing is recognized as a significant part of developing questionnaires for patient reported outcome measures (PROMs). The cognitive interviewing process used in PROM development will be adapted in this study to test the Steroid PRO in new disease populations. Cognitive interviewing will be carried out using pragmatic, light-touch interviews, underpinned by think aloud techniques and clean language principles.

SUMMARY:
Testing a questionnaire about treatment with steroids for skin, lung or gastric conditions

DETAILED DESCRIPTION:
Glucocorticoid drugs, also known as 'steroids', are used to treat a range of diseases. It is well-known that steroids can cause many unwanted side-effects. The investigators are interested in measuring the impact of steroids on quality of life, from the patients' perspective.

In a previous part of this study, the investigators interviewed participants treated with steroids for a range of rheumatic conditions. The participants were asked how taking steroids affects their everyday lives. A patient questionnaire (the 'Steroid PRO') was then created focused on the topics identified as being most important to participants.

Now the investigators would like to test this questionnaire with new participants, aged 18 or over, who are taking steroids for other conditions. This could include participants who have inflammation in the lungs, skin, or bowels. The investigators will also ask for feedback from the medical teams who care for those who have these conditions.

The study involves a single interview with a researcher, either online or by telephone. Participants who want to take part will be given information about the study and asked to give written consent. Participants will be asked to talk about the wording of the questionnaire and how relevant and feasible it is to them.

This part of the study is funded by Sanofi Research and Development. The work is being carried out by independent researchers at the University of the West of England (UWE, Bristol). Participants will be recruited from hospitals in the UK and USA.

The investigators hope that the Steroid PRO questionnaire will be used in future research trials about steroid treatment and alternatives to steroids. The Steroid PRO questionnaire could also be used in clinics to improve communication between clinicians and patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Diagnosed with an autoimmune or inflammatory respiratory, gastroenterology or dermatology condition
* Treatment with glucocorticoids with intravenous or oral glucocorticoids for an autoimmune or inflammatory condition within the previous year (or longer duration).
* Ability to give consent.

Exclusion Criteria:

* Aged <18 years old
* No autoimmune or inflammatory respiratory, gastroenterology or dermatology diagnosis
* Not treated with glucocorticoids with intravenous or oral glucocorticoids for an autoimmune or inflammatory condition within the previous year (or longer duration)
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For each of the medical specialties (respiratory, gastroenterology, dermatology), 20 patients will be purposively sampled to include a spectrum of participants with a range of different diseases and demographics (age, gender, country) for each indication.
  Key conditions will include inflammatory bowel disease (Ulcerative Colitis, Crohn's disease, Eosinophilic gastroenteritis), dermatological conditions (e.g subacute cutaneous lupus erythematosus (SCLE) systemic vasculitis, pemphigus, pemphigoid, atopic dermatitis), and respiratory conditions (asthma, COPD and interstitial lung disease).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Steroid PRO | November 2022 - May 2024
  Validated outcome measure to capture the impact of treatment with glucocorticoids on health related quality of life (Bridgewater ARD 2023). 15 item questionnaire, 4 domains (Impact on Appearance, Psychological Impact, Social impact and Treatment Concerns). Steroid PRO is the full title of the outcome measure. A PRO is a patient reported outcome. Higher scores equal greater impact on health related quality of life. Raw scores: minimum possible score 0, maximum 45.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna C Robson, FRCP PhD, Principal Investigator — University of the West of England
Locations (1):
- University of the West of England, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bridgewater S, Shepherd MA, Dawson J, Richards P, Silverthorne C, Ndosi M, Almeida C, Black RJ, Cheah JTL, Dures E, Ghosh N, Hoon EA, Lyne S, Navarro-Millan I, Pearce-Fisher D, Ruediger C, Tieu J, Yip K, Mackie SL, Goodman S, Hill C, Robson JC. Measuring the impact of steroid therapy on health-related quality of life in patients with rheumatic diseases: international development of a glucocorticoid treatment-specific patient-reported outcome measure. Rheumatology (Oxford). 2023 Nov 2;62(11):3565-3575. doi: 10.1093/rheumatology/kead081. PMID 36840642
- [Background] Bridgewater S, Ndosi M, Dawson J, Richards P, Silverthorne C, Dures E, Goodman SM, Hill C, Mackie SL, Robson JC. Validation of a new glucocorticoid-specific Patient-Reported Outcome Questionnaire (the Steroid PRO). Ann Rheum Dis. 2024 Feb 15;83(3):394-400. doi: 10.1136/ard-2023-224946. PMID 37949468
- [Derived] Sweeney AT, Bridgewater S, Orme J, Sattui SE, Sharp M, Richards P, Silverthorne CA, Arthurs E, Creed T, Osborne G, Dunhill G, Dawson J, Dures E, Barratt SL, Ramonell RP, Patton T, Goodman SM, Hill CL, Mackie SL, Ndosi M, Robson JC. Impact of glucocorticoids on patients' quality of life: a qualitative study assessing face validity and feasibility of the Steroid PRO in patients with inflammatory gastroenterology, respiratory and dermatology conditions. BMJ Open. 2025 Feb 5;15(2):e089225. doi: 10.1136/bmjopen-2024-089225. PMID 39909511